CLINICAL TRIAL: NCT04139239
Title: Diagnostic Accuracy of the Vegetative and Minimally Conscious State: Clinical Consensus Versus Standardized Neurobehavioral Assessment
Brief Title: Diagnostic Accuracy of the Vegetative and Minimally Conscious State
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Principal Investigator, Hangzhou Normal University
Other Study IDs: 2018N56745
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Disorder of Consciousness; Minimally Conscious State
Keywords: Disorders of consciousness; Coma Recovery Scale-revision; Diagnostic accuracy
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with disorders of consciousness
  Interventions: Diagnostic Test: Coma Recovery Scale-revision

INTERVENTIONS:
Diagnostic Test: Coma Recovery Scale-revision — Patients were assessed by Coma Recovery Scale-revision to detect the DOC patients enrolled by clinicians.

SUMMARY:
The aim of this study was to investigate diagnostic accuracy of the vegetative and minimally conscious state: Clinical consensus versus standardized neurobehavioral assessment

DETAILED DESCRIPTION:
In this study, DOC patients with clinical consensus of DOC were enrolled. The investigators used Coma Recovery Scale-revision (CRS-R) to assess consciousness levels for all DOC patients during ten days.

ELIGIBILITY:
Inclusion

1. at least 18 years old;
2. acquired brain injury;
3. no neuromuscular blockers or sedatives were used within 48 hours of enrollment.

Exclusion Criteria:

1. there are functional disorders caused by progressive mental diseases;
2. persistent seizures;
3. unstable vital signs;
4. double upper limb frustration, fracture.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with DOC chosen by clinician were included in the study at Department of Neurology and Rehabilitation center of hospital. All patients were diagnosed by the Coma Recovery Scale-revision (CRS-R) for five times at least within 10 days.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Assessed by the Coma Recovery Scale-Revised | Within 10 days
  All patients were assessed by the Coma Recovery Scale-Revised within 10 days to detect the consciousness level. CRS-R consists of six sub-scales with 23 items, which evaluate the patients' auditory, visual, motor, Oromotor/Verbal, communication and arousal functions. For each subscale, the lower score reflected reflexivity related to the brain stem, while the higher score reflected non-reflexivity related to higher cortical functions (0-23).

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro., Study Chair — Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Farquhar I, Fairclough JA. Sciatic block in lower limb surgery. Injury. 1990 Mar;21(2):107-9. doi: 10.1016/0020-1383(90)90066-4. PMID 2351462
- [Background] van Erp WS, Lavrijsen JC, Vos PE, Bor H, Laureys S, Koopmans RT. The vegetative state: prevalence, misdiagnosis, and treatment limitations. J Am Med Dir Assoc. 2015 Jan;16(1):85.e9-85.e14. doi: 10.1016/j.jamda.2014.10.014. PMID 25528282
- [Background] Stender J, Gosseries O, Bruno MA, Charland-Verville V, Vanhaudenhuyse A, Demertzi A, Chatelle C, Thonnard M, Thibaut A, Heine L, Soddu A, Boly M, Schnakers C, Gjedde A, Laureys S. Diagnostic precision of PET imaging and functional MRI in disorders of consciousness: a clinical validation study. Lancet. 2014 Aug 9;384(9942):514-22. doi: 10.1016/S0140-6736(14)60042-8. Epub 2014 Apr 15. PMID 24746174
- [Derived] Wang J, Hu X, Hu Z, Sun Z, Laureys S, Di H. The misdiagnosis of prolonged disorders of consciousness by a clinical consensus compared with repeated coma-recovery scale-revised assessment. BMC Neurol. 2020 Sep 12;20(1):343. doi: 10.1186/s12883-020-01924-9. PMID 32919461